CLINICAL TRIAL: NCT00629200
Title: A Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Sodium Stibogluconate in Combination With Interferon Alpha-2b for Patients With Advanced Malignancies
Brief Title: Sodium Stibogluconate With Interferon Alpha-2b for Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: VioQuest Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0354; NCI-2010-01525 (Registry Identifier: NCI CTRP); NCT01479309 (obsolete NCT alias)
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Advanced Cancer; Solid Tumors
Keywords: Advanced Malignancies; Solid Tumors; Melanoma; Renal Cell Carcinoma; Phase I Studies; Sodium Stibogluconate; Interferon Alpha-2b; Intron A; SSG
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell | interventions — Antimony Sodium Gluconate; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SSG + Intron A (Experimental): Sodium Stibogluconate (SSG) 400 mg/m^2 intravenous (IV) daily on days 1-5 + Interferon Alfa-2b (Intron A) 3x10^6 units subcutaneously three times weekly
  Interventions: Drug: Sodium Stibogluconate; Drug: Interferon Alpha-2b

INTERVENTIONS:
Drug: Sodium Stibogluconate — 400 mg/m^2 IV daily on days 1-5.
  Other Names: SSG
Drug: Interferon Alpha-2b — 3x10^6 units subcutaneously three times weekly
  Other Names: Intron A

SUMMARY:
Primary Objective:

-To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of SSG in combination with IFN alpha2b in patients with advanced malignancies.

Secondary Objectives:

* To correlate the AUC of SSG with clinical toxicity and efficacy.
* To quantify the effect of SSG on IFN alpha2b induced gene modulation and signal transduction pathways.
* To characterize the effects of SSG on PTPases SHP-1 and SHP-2.
* To assess the safety, efficacy, and PK of SSG in combination with IFN alpha2b.

DETAILED DESCRIPTION:
Sodium stibogluconate is a drug that is able to block an enzyme in the cells that is responsible for cell growth. By blocking this enzyme, it may be able to prevent cancer cells from multiplying.

Interferon alfa-2b is a drug that activates an immune response to infections in the body. By triggering an immune response, this drug may help to prevent some cancer cells from growing and multiplying. You will receive treatment with both sodium stibogluconate and interferon alfa-2b, because sodium stibogluconate may improve the effectiveness of interferon in treating the cancer.

Participants will be enrolled in groups of 3 on this study, and the doses of the study drugs will be escalated for each group. This means that each new group of 3 participants will get a higher dose of the study drugs than the group before them. This will continue until the highest tolerable dose combination is found.

Once the highest tolerable dose has been found, up to an additional 9 participants, called the expansion group, will receive study drug at that dose. Your doctor will tell you if you are in the expansion group.

If you are found to be eligible to take part in this study, you will go to the clinic to start treatment. During Cycle 1, you will be given sodium stibogluconate once a day by vein during Days 1-5. On Days 8-12, you will be given sodium stibogluconate once a day by vein, and you will be given interferon alfa-2b for 3 days by injection just under the skin on Days 8, 10, and 12. For every cycle after Cycle 1, you will be given sodium stibogluconate once a day by vein during Days 1-5 and 8-12, and you will be given interferon alfa-2b for 3 days by injection just under the skin on Days 1, 3,5, 8, 10, and 12. Treatment cycles will last about 3 weeks (2 weeks on treatment, followed by 1 week off treatment).

During each visit to the clinic, you will be asked how you are feeling, and your vital signs will be measured. You will have a complete physical exam the first day of every cycle. On Days 1, 8, and 12 of every cycle, you will have a urine test to check the function of your kidneys, and blood (about 3 teaspoons) will be drawn for routine tests. On Days 1, 8, and 12 of every cycle and during your last study visit, you will have an additional blood draw (about 5 teaspoons) for immunological testing (to help researchers learn how your body fights disease) before treatment. On Days 1, 5, 8, and 12 of every cycle, you will have an ECG after you receive treatment.

At some time during the week before Day 1 of Cycle 1 and on Day 12 of Cycle 2, you may have a tumor biopsy to check the status of the disease before you receive the study drug. To perform a tumor biopsy, the affected area is numbed with anesthetic, and a small amount of tumor tissue is withdrawn through a large needle. Your doctor will tell you if this may be necessary.

On Days 1, 2, 9, 12, and 13 of Cycle 1, you will have blood drawn (about 1 teaspoon each) for PK testing. On Days 1, 8, and 12, the PK testing will be done before, 30 minutes after, and 2 hours after you receive the study drug. On Days 2 and 9, the PK testing will be done before treatment. On Day 13, the PK testing will be done 24 hours after you received treatment on Day 12.

After Cycle 1, you will be scheduled to return to the clinic in 10 days to receive treatment for Cycle 2, which will follow in the same manner as Cycle 1.

At the end of Cycle 2 and every even-numbered cycle (Cycles 4, 6, 8, and so on) after that, you will have imaging studies, such as x-rays and CT scans, to check the status of your tumors.

If the disease does not get worse and you do not experience any intolerable side effects after Cycle 1, you will continue on to Cycle 2, and so on. If at any time the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

This is an investigational study. Sodium stibogluconate is not FDA approved or commercially available. It is authorized for use in research only. Interferon alfa-2b is approved by the FDA for the treatment of some types of cancers (solid tumors). The combination of these drugs is investigational in this study. Their use together is authorized for use in research only.

However, if sodium stibogluconate becomes commercially available while you are still on study. Up to 54 patients will take part in this multicenter study. Up to 35 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign a written informed consent document and are able to comply with the study protocol for the duration of the study.
2. Patients who have a histologically or cytologically confirmed diagnosis malignancy (patients with measurable or non-measurable disease) who have progressed following effective therapy or for which no effective therapy exists.
3. Patients who are greater than or equal to 18 years of age.
4. Patients who have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
5. Patients who have an estimated life expectancy of 3 months.
6. Patients who have a normal cardiac ejection fraction, >50% estimated by 2 D Echocardiogram or MUGA.
7. Patients who have adequate organ function as indicated by the following laboratory values obtained within 10 days prior to the first dose of SSG: Granulocytes>/=1,500 microliter, Platelets>/= 100,000 microliter, Hemoglobin >/=9.0 g/dL,Creatinine (Cr) </= 1.5 mg/dL, Bilirubin Normal limits, or <2.0 x ULN with liver metastases, Aspartate aminotransferase (AST) <2.5 * ULN or <5.0 * ULN with liver metastases, Alanine aminotransferase (ALT)<2.5 * ULN or <5.0 * ULN with liver metastases.

Exclusion Criteria:

1. Patients on concurrent immunotherapy, including IFN therapy (prior therapy is allowed if >/= 4 months since immunotherapy).
2. Patients who have received investigational drugs including immunotherapy, gene therapy, hormone therapy, biologic therapy, radiation therapy, chemotherapy, or had major surgery within 3 weeks of study enrollment
3. Patients who have not recovered from acute toxicity of previous therapy prior to enrollment.
4. Patients with medically uncontrolled cardiovascular illness, unstable angina, congestive heart failure, history of myocardial infarction, electrocardiogram (ECG) abnormalities suggestive of cardiac conduction delay (QTc >0.47 seconds), history of atrial fibrillation or flutter, or other serious clinically significant cardiac arrhythmia
5. Patients who have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant.
6. Pregnant or lactating women, and fertile women or men unless surgically sterile or using effective contraception; All female patients of childbearing potential or < 1 year postmenopausal must have a negative beta human chorionic gonadotropin (βhCG) pregnancy test at baseline and be practicing a medically acceptable method of birth control (oral contraceptives for at least 3 months, implantation of an intrauterine device at least 2 months, or barrier methods [e.g. vaginal diaphragm, vaginal sponge, or condom with spermicidal jelly]). These must be continued for 3 months after study initiation
7. Patients who use daily glucocorticoids except for physiological replacement.
8. Patients who are known to be positive for Hepatitis B surface antigen, Hepatitis C or human immunodeficiency virus (HIV).
9. Patients with prior history of solid organ allografts or allogeneic bone marrow transplant.
10. Patients who have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
11. Patients who have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Patient who have symptomatic or untreated central nervous system metastases.
13. Patients taking the following medications will not be eligible: Amiodarone (Cordarone); Disopyramide (Norpace); Dofetilide (Tikosyn); Procainamide (Procanbid, Pronestyl); Quinidine (Quinaglute); Sotalol (Betapace); Erythromycin; Azithromycin (Z-pack), cont'd
14. Clarithromycin (Biaxin); Pentamidine (Pentacarinat); Trimethoprim-sulfamethoxazole (Bactrim); Bepridil (Vascor); Phenothiazines-prochlorperazine (Compazine), promethazine (Phenergan), chlorpromazine (Thorazine) or any antipsychotic medication; Butyrophenones-Haloperidol (Haldol), cont'd
15. Risperidone (Risperdal); Tricyclic or tetracyclic antidepressants-imipramine (Tofranil), amitriptyline (Elavil), desipramine (Norpramin), nortriptyline (Pamelor); Monoamine oxidase inhibitors; High dose methadone; Arsenic trioxide; Dolasetron (Anzemet); Any herbal preparations; or • Chronic need for colony stimulating factors (i.e., GM-CSF), erythropoietin use is permitted.
16. Patients with a history of hypersensitivity to IFN a-2b or SSG or any of their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-09-13 (Actual); Primary Completion 2010-02-10 (Actual); Study Completion 2010-02-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of SSG in combination with IFN alpha2b | Continuous assessment with each 3 week cycle
  MTD defined as the highest dose at which no dose limiting toxicity (DLT) occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - U.T.M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org